CLINICAL TRIAL: NCT05653856
Title: A Multi-Center, Open-Label, Randomized Phase 2 Study of Copper Cu 64 PSMA I&T Injection in Patients With Histologically Proven Metastatic Prostate Cancer
Brief Title: Cu-64-PSMA-I&T Positron Emission Tomography (PET) Imaging of Metastatic PSMA Positive Lesions in Men With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Curium US LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CURCu64PSM0001 (Phase II)
Record Dates: First submitted 2022-11-07; First posted 2022-12-16 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Metastasis From Malignant Tumor of Prostate (Disorder)
Keywords: PSMA; Prostate Cancer; PET; SOLAR; Cu-64 PSMA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic Imaging with 64Cu-PSMA-I&T (Experimental): 64Cu-PSMA I&T
  Interventions: Drug: 64Cu-PSMA I&T

INTERVENTIONS:
Drug: 64Cu-PSMA I&T — Radiolabeled Receptor-Targeted Diagnostic Product

SUMMARY:
This is a prospective, open-label Phase 2 study to evaluate copper Cu 64 PSMA I&T injection for PET/CT imaging in patients with recurrent metastatic prostate cancer after radical prostatectomy or radiation therapy.

DETAILED DESCRIPTION:
The study will include a group of 26 patients with metastatic prostate cancer. Each patient will be administered a 7-9 mCi intravenous dose of copper Cu 64 PSMA I&T injection. PET/CT images will be acquired for all patients at 1 hour ± 15 minutes and 4 hours ± 30 minutes post copper Cu 64 PSMA I&T injection.

The PET/CT images will be interpreted independently by three readers blinded to all patient information. Each patient study will be assessed and scored for the detection of prostate cancer. Specifically, each reader will categorize images as "Disease" or "No Disease" based only on tumor uptake of copper Cu 64 PSMA-I&T in each of the four regions: 1) prostate bed or prostate gland, 2) lymph nodes (pelvic and extra pelvic), 3) bone, and 4) viscera/soft tissue. Analysis of the reads will be used for determination of the CLR and CDR for 1 hour and 4-hour post-injection imaging of copper Cu 64 PSMA I&T PET/CT by comparison to the Composite Reference Standard.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven prostate adenocarcinoma.
2. Prior radical prostatectomy or radiation therapy with curative intent.
3. Recurrence of disease defined as:

   1. Prior Radical Prostatectomy: PSA > 0.2 ng/mL, or
   2. Prior Radiation Therapy: 2 ng/mL rise in PSA over post-treatment nadir
4. Patients with at least one extraprostatic site of disease suspected based on prior imaging or diagnosed by biopsy.
5. Age greater than or equal to 18 years.
6. Able to understand and provide signed written informed consent.

Exclusion Criteria:

1. Androgen deprivation therapy (ADT) or other therapies targeting the androgen pathway, unless subject has a rising PSA level.
2. Body weight greater than 350 lb (158 kg).
3. Investigational therapy within the past 30 days.
4. Creatinine clearance (ClCr) less than 30 mL/min.
5. Participants who are capable of fathering a child and who are unwilling to take precautions to prevent pregnancy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Yale University, New Haven, Connecticut
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Saint Louis University, St Louis, Missouri
  - John J. Cochran Veterans Hospital, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - XCancer Omaha/Urology Cancer Center, Omaha, Nebraska
  - MD Anderson, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 9 sites across USA, Recruitment was initiated on 30 November, 2022 and was closed on 17 May 2023.
Period: Overall Study
Arm/Group | Diagnostic Imaging With 64Cu-PSMA-I&T
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic Imaging With 64Cu-PSMA-I&T
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: CM] — centimeters (cm)
  CM | 176.0 (6.45)
Weight [Mean (Standard Deviation); unit: KG] — kilograms (kg)
  KG | 91.3 (15.87)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.43 (4.544)

OUTCOME MEASURES:

1. Primary Outcome: Region-Level Correct Localization Rate (CLR)
Description: To determine the region-level correct localization rate (CLR) of copper Cu 64 PSMA I&T injection PET/CT imaging for the detection of recurrent metastatic prostate cancer at 1 hour and 4 hours post injection. The CLR is defined as the percentage of regions containing at least one true PET positive lesion, with exactly localized correspondence between PET/CT imaging and the Composite Reference Standard regardless of any co-existent false positive findings, within the same region, out of all regions containing at least one PET positive finding.
Time Frame: 4 Hours
Population: The PET/CT images were acquired for all 26 patients at 1 hour and 4 hours post copper Cu 64 PSMA I&T injection and interpreted independently by 3 readers blinded to clinical information and findings on the composite reference standard.
Measure: Mean (95% Confidence Interval); unit: percentage of Regions
Arm/Group | Diagnostic Imaging With 64Cu-PSMA-I&T
Number analyzed (Participants) | 26
percentage of Regions
  Reader 1 (1-Hour Image) | 86.67 [69.28 to 96.24]
  Reader 1 (4-Hour Image) | 86.67 [69.28 to 96.24]
  Reader 2 (1-Hour Image) | 76.67 [57.72 to 90.07]
  Reader 2 (4-Hour Image) | 80.00 [61.43 to 92.29]
  Reader 3 (1-Hour Image) | 80.00 [61.43 to 92.29]
  Reader 3 (4-Hour Image) | 80.00 [61.43 to 92.29]

2. Primary Outcome: Patient-Level Correct Detection Rate (CDR)
Description: To determine the patient-level correct detection rate (CDR) of copper Cu 64 PSMA I&T injection PET/CT imaging for the detection of recurrent metastatic prostate cancer at 1 hour and 4 hours post injection. The CDR is defined as the percentage of patients who have at least one true PET positive lesion, with exactly localized correspondence between PET imaging and the Composite Reference Standard, regardless of any co-existent false positive findings, out of all patients who are scanned.
Time Frame: 4 Hours
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of Patients
Arm/Group | Diagnostic Imaging With 64Cu-PSMA-I&T
Number analyzed (Participants) | 26
percentage of Patients
  Reader 1 (1-Hour Image) | 84.21 [68.04 to 100.00]
  Reader 1 (4-Hour Image) | 84.21 [68.04 to 100.00]
  Reader 2 (1-Hour Image) | 77.19 [58.79 to 95.59]
  Reader 2 (4-Hour Image) | 79.82 [61.55 to 98.10]
  Reader 3 (1-Hour Image) | 80.70 [63.71 to 97.69]
  Reader 3 (4-Hour Image) | 80.70 [63.71 to 97.69]

3. Primary Outcome: Incidence of Adverse Events
Description: Adverse events (AEs) were assessed from the time of copper Cu 64 PSMA I&T injection throughout the24-hour assessment period. AEs were assessed and graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: 24 Hours
Population: All 26 patients were analyzed for Adverse Events through the monitoring of clinical and laboratory safety parameters.
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic Imaging With 64Cu-PSMA-I&T
Number analyzed (Participants) | 26
Participants
  Adverse Events (AEs) | 3
  Serious Adverse Events (SAEs) | 0

4. Secondary Outcome: Score of Image Quality
Description: To compare the diagnostic quality of PET/CT images obtained at 1 hour and 4 hours post copper Cu 64 PSMA I&T injection. Image quality score is based on a scale of 0-2 where 0 is not of diagnostic quality and 2 is of best diagnostic quality.
Time Frame: 4 Hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic Imaging With 64Cu-PSMA-I&T
Number analyzed (Participants) | 26
Participants
  Reader 1 (1-Hour Post Dose): Inadequate | 0
  Reader 1 (1-Hour Post Dose): Questionable | 0
  Reader 1 (1-Hour Post Dose): Acceptable | 26
  Reader 1 (4-Hour Post Dose): Inadequate | 0
  Reader 1 (4-Hour Post Dose): Questionable | 0
  Reader 1 (4-Hour Post Dose): Acceptable | 26
  Reader 2 (1-Hour Post Dose): Inadequate | 0
  Reader 2 (1-Hour Post Dose): Questionable | 2
  Reader 2 (1-Hour Post Dose): Acceptable | 24
  Reader 2 (4-Hour Post Dose): Inadequate | 0
  Reader 2 (4-Hour Post Dose): Questionable | 0
  Reader 2 (4-Hour Post Dose): Acceptable | 26
  Reader 3 (1-Hour Post Dose): Inadequate | 0
  Reader 3 (1-Hour Post Dose): Questionable | 0
  Reader 3 (1-Hour Post Dose): Acceptable | 26
  Reader 3 (4-Hour Post Dose): Inadequate | 0
  Reader 3 (4-Hour Post Dose): Questionable | 0
  Reader 3 (4-Hour Post Dose): Acceptable | 26

ADVERSE EVENTS:
Time Frame: 24 Hours
Arm/Group | Diagnostic Imaging With 64Cu-PSMA-I&T
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period no less than 90 days but less than or equal to 120 days from the time submitted to the sponsor for review. Also, the PI can utilize results of clinical tests and site and patient outcome information only for its own internal non-commercial teaching, research, patient care, and treatment and publication purposes.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT05653856/Prot_SAP_000.pdf